CLINICAL TRIAL: NCT05620927
Title: Clinical Factors Determining the Occurrence of Impaired Awareness of Hypoglycemia (IAH) in Adult Patients With Type 1 Diabetes
Brief Title: Hypoglycemia Awareness Study in Diabetes Type 1
Acronym: HAD-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aleksandra Araszkiewicz, Professor, Poznan University of Medical Sciences
Other Study IDs: 795/22
Record Dates: First submitted 2022-11-06; First posted 2022-11-17 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Type 1 Diabetes; Hypoglycemia Unawareness; Cardiac Autonomic Neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — venous blood smple: A1c, lipids, creatinine, TSH, cortisol urine: albumine / creatinine ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 1 diabetes: Type 1 diabetes > 10 years duration of diabetes

SUMMARY:
The goal of this observational study is to assess clinical factors associated with the occurrence of impaired hypoglycemia awareness in adult patients with type 1 diabetes

The main questions it aims to answer are:

1. Determination of the prevalence of impaired hypoglycemia awareness (IAH) in adult patients with type 1 diabetes in the Polish population.
2. Assessment of the clinical usefulness of commonly used standardized scales for the assessment of IAH.
3. Determination of the clinical factors associated with the occurrence of impaired hypoglycemia awareness in adult patients with type 1 diabetes.
4. Determination of the relationship between the occurrence of IAH and the diagnosis of cardiac autonomic neuropathy.
5. Determination of the relationship between impaired hypoglycemia awareness in adult patients with type 1 diabetes and the occurrence of cognitive impairment.

Participants will:

* fill the standard questionnaires regarding hypoglycemia awareness: Gold, Clarck, HypoA-Q.
* have late complications of diabetes checked
* have procedure of cardiac autonomic neuropathy assessment
* have standard laboratory evaluation during hospitalization

DETAILED DESCRIPTION:
Hypoglycemia defined as a blood glucose level ≤70 mg / dL is the most common acute complication in patients with type 1 diabetes (T1D). Hypoglycemia is accompanied by alarm symptoms caused by neuroglycopenia and stimulation of the autonomic nervous system caused by the response of counterregulatory hormones. Being aware of the symptoms of hypoglycemia helps patients to recognize hypoglycemia and begin self-treatment. In people experiencing recurrent episodes of hypoglycemia, the counter-regulatory hormonal response may be abnormal, reducing the perception of hypoglycemia. This condition is called impaired awareness of hypoglycemia (IAH) and affects up to 40% of T1D patients. IAH is the reduction or loss of the ability to recognize low blood glucose and respond correctly to the onset of hypoglycemia. It is a significant clinical problem among patients with T1D. IAH exposes patients to severe hypoglycemia, which is associated with impaired consciousness and damage to nerve cells. Therefore, patients with T1D with IAH may feel fear of developing hypoglycemia, which often results in a lack of compliance with the rules of insulin therapy, and thus difficulties in achieving good glycemic control. This can result in chronic hyperglycemia and the development of microvascular and macrovascular complications.

Common episodes of hypoglycemia can lead to disturbances in the development and maturation of neurons, resulting in cognitive impairment, structural changes in the central nervous system, lower levels of intellectual abilities, and behavioral disturbances. MRI studies in patients with T1D and IAH showed brain changes including gray matter and white matter. These changes correlate with the frequency of severe hypoglycemia and, in some areas of the brain, with the severity of IAH.

Hypoglycemia unawareness may also be due to the presence of diabetic cardiovascular autonomic neuropathy (CAN). CAN is an established factor associated with severe hypoglycemia. By reducing the catecholamine counter-regulatory response to hypoglycemia as well as the severity of autonomic warning symptoms, CAN may contribute to IAH. The American Diabetes Association (ADA) recommends screening for CAN in patients with impaired hypoglycemia awareness. However, the relationship between CAN and IAH has not been well established. Few data suggested CAN as a possible cause of IAH, however, further studies in patients with T1D ruled out the association of CAN with IAH. Olsen et al. assessed the relationship of IAH with the presence of CAN and peripheral neuropathy in a group of 66 patients with a 31-year history of T1D. The study showed that adults with IAH compared to the control group (adults with T1D without IAH) did not differ in the incidence of CAN and peripheral neuropathy. Paes et al. in the group of 98 patients with a 13-year duration of CT1 also observed no difference in the incidence of CAN among patients with IAH compared to those with T1D without IAH. However, they confirmed the relationship between age, diabetes duration, number of severe hypoglycemic episodes, and creatinine clearance with IAH. Patients with IAH had a longer T1D duration and lower creatinine clearance compared to the control group. Moreover, in people with impaired hypoglycemia awareness, the number of severe hypoglycemia episodes was higher compared to those with normal hypoglycemia.

A simple and widely used method of assessing hypoglycemia awareness is the use of validated questionnaires in which patients report specific situations in their life related to hypoglycemia. Four questionnaires are known to diagnose awareness of hypoglycemia: Gold, Clarke, Pedersen-Bjergaard, and HypoA-Q. The advantage of using the above-mentioned questionnaires as a method of assessing hypoglycemia awareness is non-invasiveness, no / minimal cost, reporting experiences from actual episodes of hypoglycemia, the possibility of use in large patient populations, and the possibility of clinical application.

Identifying the factors that influence IAH could help draw attention to patients at risk of its consequences. Then, they could undergo hypoglycemia training, education to optimize insulin dosing, or stricter control, e.g. thanks to the use of continuous glucose monitoring systems.

Methods:

Observational, single-center study

1. Inclusion of 245 consecutive patients (women and men over 18 years of age) with type 1 diabetes, with disease duration> 10 years, hospitalized at the Department of Internal Medicine and Diabetology, Poznan University of Medical Sciences
2. Assessment of the level of hypoglycemia awareness using standardized questionnaires: HYPOA-Q, Clarke, Gold. These are the three most commonly used scales for assessing the IAH. The endpoint, i.e. impaired hypoglycemic awareness, will be any abnormal result in one of the following scales indicating IAH (HYPOA-Q score above the median in the study population, Gold and Clarke ≥ 4)
3. Evaluated factors from the history - age, duration of diabetes, smoking, physical activity, number of severe hypoglycemia and diabetic ketoacidosis in life, partial clinical remission after diagnosis of diabetes, presence of comorbidities (hypertension, hypercholesterolemia), number of hours of sleep, shift work, method of insulin therapy used by the patient, A1c values from the history of the last 5 years.
4. Assessment of glycemic control from reports from continuous glucose monitoring systems and glucometers - number of hypoglycemic episodes <54 and ≤70 mg / dL in the last 4 weeks (meter reading) or duration of hypoglycemia, mean glycemia and parameters of glucose variability
5. Daily dose of insulin
6. Anthropometric measurements: body weight, height, waist and hip circumference, body weight composition
7. Laboratory tests: performed on an empty stomach, collecting about 8 ml of venous blood and a urine sample of 50-100 ml. These are tests routinely performed in the hospital to assess metabolic control in type 1 diabetes.
8. Study of the accumulation of advanced glycation products in tissues based on the level of skin autofluorescence
9. Montreal Cognitive Assessment Scale - a tool for screening the assessment of mild cognitive impairment. The 10-minute test allows you to assess attention and concentration, executive functions, memory, language, visual and spatial functions, conceptual thinking, calculation skills and orientation. The maximum number of points that can be obtained is 30. A score below 26 points suggests a cognitive impairment.
10. Hypoglycemia Fear Survey - questionnaire assessing fear of hypoglycemia in the last four weeks.
11. Tests for the presence of chronic complications of diabetes mellitus: diabetic retinopathy, diabetic kidney disease, peripheral neuropathy, and cardiovascular autonomic neuropathy:

Expected results:

1. In the opinion of experts, the prevalence of IAH in the Polish population in adult patients with type 1 diabetes with disease duration over 10 years is estimated at least 20%. We assume N = (the literature says that there may be about 3.5 million diabetic patients in Poland, of which about 10% is DM1), therefore N = 35,000, then I assume that the fraction p = 20% and the significance level p = 0.05 and the permissible estimation error e = 5%, therefore the minimum necessary number is n = 245.
2. The scales used to assess IAH have different clinical utilities. The HYPOA-Q scale allows us to recognize the problem of IAH in more patients (higher sensitivity).
3. Determination of clinical factors independently related to the incidence of IAH. Expected independent factors related to IAH are age, disease duration, lifetime number of severe hypoglycemia and diabetic ketoacidosis, duration of hypoglycemia or number of hypoglycemia in the last 4 weeks, and macroangiopathy.
4. Determination of the relationship between the occurrence of IAH and the diagnosis of cardiac autonomic neuropathy. Expected confirmation of the existence of such a relationship.
5. Confirmation of the relationship between impaired hypoglycemia awareness in adult patients with type 1 diabetes and the occurrence of cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Duration of diabetes > 10 years
* Consent to participate in the study

Exclusion Criteria:

* Age under 18
* Duration of diabetes> 10 years
* Neurodegenerative diseases (Parkinson's disease, Alzheimer's disease, Huntington's disease)
* Multiple sclerosis
* Mental disorders
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Impaired awareness of hypoglycemia (IAH) - HypoA-Q | one year
  Determination of the prevalence of impaired hypoglycemia awareness (IAH) in adult patients with type 1 diabetes in the Polish population in % in the study population measured by the HypoA-Q.
Impaired awareness of hypoglycemia (IAH) - Gold Questionnaire | one year
  Determination of the prevalence of impaired hypoglycemia awareness (IAH) in adult patients with type 1 diabetes in the Polish population in % in the study population measured by the Gold scale.
  Gold Questionnaire contains one question asking individuals to report their experience of detecting hypoglycemic events with a score ranging from 1 (always aware) to 7 (never aware) on the Likert scale.
Impaired awareness of hypoglycemia (IAH) - Clarke's Questionnaire | one year
  Determination of the prevalence of impaired hypoglycemia awareness (IAH) in adult patients with type 1 diabetes in the Polish population in % in the study population measured by the Clarke's Questionnaire - Consists of eight questions assessing the prior experience of hypoglycemia, such as a history of severe hypoglycemia development and blood glucose levels at which patients begin to detect symptoms of hypoglycemia. The questionnaire generates a score (0-7) based on the patient's responses.

SECONDARY OUTCOMES:
diagnosis of cardiac autonomic neuropathy. | one year
  measurement of heart rate variability using the CARDIOSYS EXTRA system (MDE GmbH). It is a non-invasive method. The patient's heart rate variability under the influence of certain standardized stimuli is tested (supine test, deep breathing test, Valsalva maneuver, orthostatic test, hand grip test). During the examination, the ECG of the examined person is monitored on the computer screen. The program recognizes R waves and calculates successive R-R intervals and their variability. Based on the calculated differences in R-R intervals, specific parameters for the assessment of autonomic neuropathy are calculated and compared with the norm values for age and gender. Autonomic neuropathy is diagnosed if two of the four tests are abnormal
Hypoglycemia Fear Survey | one year
  HFS-II questionnaire (Hypoglycemia Fear Survey) - questionnaire assessing fear of hypoglycemia in the last four weeks. It consists of two subscales. The first: Behavior contains 15 questions about what to do to avoid low blood glucose and its consequences. Second: Concerns includes 18 questions about concerns about low blood glucose levels. For each question, the patient scores between 0 (never) and 4 (almost always). The results are the sum of points separately for each subscale. The higher the score, the greater the fear of hypoglycemia.
occurrence of cognitive impairment | one year
  MOCA Questionnaire - Montreal Cognitive Assessment Scale - a tool for screening the assessment of mild cognitive impairment. The 10-minute test allows you to assess attention and concentration, executive functions, memory, language, visual and spatial functions, conceptual thinking, calculation skills and orientation. The maximum number of points that can be obtained is 30. A score below 26 points suggests a cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Araszkiewicz, Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No